CLINICAL TRIAL: NCT04758234
Title: A Randomized, Double-Blind, Single-Ascending Dose and Multiple-Dose, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3549492 in Healthy Subjects
Brief Title: A Study of LY3549492 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18082; J3H-MC-GZNA (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-02-16; First posted 2021-02-17 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LY3549492 (Part A) (Experimental): LY3549492 administered orally as single ascending doses.
  Interventions: Drug: LY3549492
- LY3549492 (Part B) (Experimental): LY3549492 administered orally as multiple ascending doses.
  Interventions: Drug: LY3549492
- Placebo (Placebo Comparator): Placebo administered orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3549492 — Administered orally.
  Arms: LY3549492 (Part A); LY3549492 (Part B)
Drug: Placebo — Administered orally.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of LY3549492 in healthy participants. The blood tests will be performed to check how much LY3549492 gets into the bloodstream and how the body handles LY3549492. This study includes two parts and will last up to approximately 76 days for each participant, including screening.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Males and females (excluding women of childbearing potential at the time of signing the informed consent)
* Glycated hemoglobin (HbA1c) value of <6.5% at screening
* Body mass index (BMI) within the range 20 to 40 kilograms per square meter (kg/m²), inclusive
* Capable of giving signed informed consent form (ICF)

Exclusion Criteria:

* Have obesity induced by endocrine disorders such as Cushing's syndrome or Prader-Willi syndrome.
* Have significant history of or current cardiovascular, respiratory, hepatic, renal, Gastro-intestine (GI) (including cholecystectomy with no sequelae, GI disease that significantly impact gastric emptying or motility, such as severe gastroparesis or pyloric stenosis even if treated), endocrine, hematological, psychiatric or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data.
* Have undergone any form of bariatric surgery.
* Have a history or presence of pancreatitis (history of chronic pancreatitis or idiopathic acute pancreatitis), elevation in serum amylase or lipase (>2.5 fold the upper limit of normal (ULN)).
* Have a personal or family history of medullary thyroid carcinoma or have Multiple Endocrine Neoplasia Syndrome Type 2.
* Have a serum calcitonin level of ≥20 nanogram/liter (ng/L) at screening, if estimated glomerular filtration rate is ≥60 milliliter/minute/1.73 square meter (mL/min/1.73 m2).
* Have an active or history of malignancy within 5 years prior to screening, except for basal cell or squamous epithelial carcinomas of the skin or in situ carcinoma of the uterine cervix that have been resected with no evidence or recurrence or metastatic disease for at least 3 years.
* Have known liver disease, obvious clinical signs, or symptoms of liver disease, acute or chronic hepatitis, or have elevations in aminotransferases (alanine aminotransferase [ALT] and aspartate aminotransferase [AST]) greater than 2 times [ULN]).
* Have total bilirubin level (TBL) >1.5 × ULN (except for participants diagnosed with Gilbert's syndrome).
* Have serum triglyceride >500 milligram/deciliter (mg/dL) at screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through final follow-up at approximately Day 76
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY3549492 | Predose up to 48 days postdose
  PK: AUC of LY3549492
PK: Maximum Concentration (Cmax) of LY3549492 | Predose up to 48 days postdose
  PK: Cmax of LY3549492

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No